CLINICAL TRIAL: NCT03166527
Title: Prospective, Open-Label, Phase IIIb Study Evaluating the Safety, Tolerability and Efficacy of Panzyga® in Patients With Chronic Inflammatory Demyelinating Polyneuropathy Administered at Standard and High Infusion Rates
Brief Title: Panzyga in CIDP Administered at Different Infusion Rates
Acronym: Panzyga-CIDP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vera Bril (Other)
Responsible Party: Sponsor-Investigator, Vera Bril, MD, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1001
Record Dates: First submitted 2017-05-08; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Immunoglobulins

STUDY DESIGN:
Intervention Model Description: Each patient with active CIDP will receive Panzyga (immune globulin) at standard and high infusion rates and will act as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label study (Other): open label study using Panzyga immune globulin 10% intravenous solution with no placebo.
  Interventions: Drug: Immune Globulin 10% Intravenous Solution

INTERVENTIONS:
Drug: Immune Globulin 10% Intravenous Solution — standard Immune lobulin 10% intravenous solution infusion at standard and high infusion rates.
  Other Names: Panzyga IVIG

SUMMARY:
Chronic inflammatory demyelinating polyneuropathy (CIDP) is a treatable form of peripheral neuropathy with suspected autoimmune cause. The current first-line treatment is IVIG (immune globulin), which is infused in a set regimen that requires 4-5 hours in a hospital day unit, taking up resources such as nursing time and hospital space. Chronic treatment is required in most cases.

DETAILED DESCRIPTION:
The proposed trial will be an exploratory, open-label, single-centre, phase IIIb safety, tolerability and efficacy study, wherein each patient acts as their own control. The primary outcome measure is safety and tolerability of panzyga in patients with active CIDP at standard and high infusion rates as measured by:

* Occurrence of all adverse events with focus on adverse drug reactions (ADRs)
* The secondary outcomes include: Patients' treatment satisfaction, proportion of patients successfully achieving higher infusion rates, health utilities associated with treatment, proportion of responders to treatment based on change in clinical scores, grip strength, and quality of life measures. The total sample size is 25-30 patients, based on a difference of 30% in adverse events rates between the standard infusion rate and the maximum rate tolerated by each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of definite or probable CIDP according to the EFNS/PNS Guideline 2010; including patients with Multifocal Acquired Demyelinating Sensory And Motor Neuropathy (MADSAM) or pure motor CIDP
2. Patients with active disease, i.e. not being in remission.
3. IVIG naïve patients with clinical indication for IVIG based on progressive or relapsing disease and adjusted INCAT (ONLS) disability score between 2 and 9 (with a score of 2 coming exclusively from leg disability).
4. Patients already receiving IVIG must be on 3- or 4-weekly IVIG treatment schedule with a calculated monthly dosage between 0.8 g/kg and 2.0 g/kg BW
5. ≥ 18 years of age
6. Voluntarily given, fully informed written consent obtained from patient before any study-related procedures are conducted
7. For enrolment into the Second Phase: At each of the last three infusions in the First Phase, administration of panzyga® had to be at the maximum infusion rate of 0.08 mL/kg/min and good tolerated- assessment by Investigator according to local site practice

Exclusion Criteria:

1. MMN with conduction block
2. Patients who previously failed immunoglobulin therapy
3. Treatment with immunomodulatory/suppressive agents (cyclosporin, methotrexate, mitoxantrone, mycophenolate mofetil or azathioprine) during the six months prior to baseline visit
4. Patients on or treated with rituximab, alemtuzumab, cyclophosphamide, or other intensive chemotherapeutic regimens, previous lymphoid irradiation or stem cell transplantation during the 12 months prior to baseline visit
5. Respiratory impairment requiring mechanical ventilation
6. Myelopathy or evidence of central nervous system demyelination or significant persisting neurological deficits from stroke, or central nervous system (CNS) trauma
7. Clinical evidence of peripheral neuropathy from another cause such as

   1. connective tissue disease or systemic lupus erythematosus (SLE)
   2. HIV infection, hepatitis, Lyme disease
   3. cancer (with the exception of basal cell skin cancer)
   4. IgM paraproteinemia with anti-myelin associated glycoprotein antibodies
8. Diabetic neuropathy
9. Cardiac insufficiency (New York Heart Association [NYHA] III/IV), cardiomyopathy, significant cardiac dysrhythmia requiring treatment, unstable or advanced ischemic heart disease
10. Severe liver disease (ALAT 3x > normal value)
11. Severe kidney disease (creatinine 1.5x > normal value)
12. Hepatitis B, hepatitis C or HIV infection
13. Thromboembolic events: patients with a history of deep vein thrombosis (DVT) within the last year prior to baseline visit or pulmonary embolism ever; patients with susceptibility to embolism or DVT
14. Body mass index (BMI) ≥40 kg/m2
15. Selective IgA deficiency with known anti-IgA antibodies
16. History of hypersensitivity, anaphylaxis or severe systemic response to immuno-globulin, blood or plasma derived products, or any component of panzyga®
17. Known blood hyperviscosity, or other hypercoagulable states
18. Use of other blood or plasma-derived products within three months prior to enrolment
19. Patients with a past or present history of drug abuse or alcohol abuse within the preceding five years prior to baseline visit
20. Patients unable or unwilling to understand or comply with the study protocol
21. Participation in another interventional clinical study with IMP treatment currently or during the three months prior to enrolment
22. Women who are breast feeding, pregnant, or planning to become pregnant, or are unwilling to use an effective birth control method (such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner) while on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-12-15 (Estimated); Study Completion 2018-12-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of all adverse events with focus on adverse drug reactions (ADRs) | 2 years
  adverse drug reactions

SECONDARY OUTCOMES:
treatment satisfaction | 2 years
  completion of questionnaire
proportion of patients successfully achieving higher infusion rates | 2 years
  descriptive analysis of number of patients
health utilities | 2 years
  completion of questionnaire
proportion of responders to treatment based on change in clinical scores | 2 years
  completion of scale
grip strength | 2 years
  measurements in kPa
quality of life measures | 2 years
  completion of scale

CONTACTS AND LOCATIONS:
Locations (1):
- UHNToronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No